CLINICAL TRIAL: NCT02966886
Title: Comparison of Shoulder Arthroplasty Techniques in the Treatment of Glenohumeral Osteoarthritis: Protocol
Brief Title: TSA Techniques in Glenohumeral OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20160779-01H
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Shoulder
Keywords: Surgical Management
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with 10-15 degrees of glenoid retroversion (Active Comparator)
  Interventions: Procedure: Eccentric Reaming; Procedure: Augmented Glenoid Component Implantation
- Participants with >15 degrees of glenoid retroversion (Active Comparator)
  Interventions: Procedure: Augmented Glenoid Component Implantation; Procedure: Posterior Glenoid Bone Grafting

INTERVENTIONS:
Procedure: Eccentric Reaming — Pre-operative CT imaging and surgical planning software based on pre-operative CT scans will be used in each case to determine the degree of eccentric ("high side") anterior reaming to within < 10 degrees of neutral glenoid version.
  Arms: Participants with 10-15 degrees of glenoid retroversion
Procedure: Augmented Glenoid Component Implantation — Patients will undergo standard glenoid preparation and implantation of a posteriorly augmented glenoid component. The degree of posterior augment will be based on pre-operative CT scan assessment and templating software with the goal of correcting glenoid retroversion to within 10 degrees of neutral version.
Procedure: Posterior Glenoid Bone Grafting — Patient will undergo a total shoulder arthroplasty as per standard technique. Glenoid version will be restored to within 10 degrees of neutral with a posterior glenoid bone graft. The bone graft will be harvested from the humeral head and fixed to the posterior glenoid with mini-fragment screws.
  Arms: Participants with >15 degrees of glenoid retroversion

SUMMARY:
Osteoarthritis (OA) of the shoulder is a disease resulting from the wearing down of cartilage over time. OA can produce pain and dysfunction at the affected joint and is a growing occurrence in an aging population. Total shoulder arthroplasty (TSA) is a surgical treatment used to treat patients with shoulder OA which involves replacing the worn-out ball and socket shoulder joint with prosthetic components. TSA is performed today with high success rates, however, complication rates associated with TSA remain prevalent particularly when the arthritis is associated with bone erosion on the glenoid (socket).

Given the high rate of revisions associated with TSA treatment in the setting of glenoid bone erosion, a number of surgical strategies have been developed. These surgical techniques include eccentric reaming which involves removing bone from the front of the socket, augmented glenoid component implantation, and posterior bone grafting to compensate for glenoid bone loss, and reverse shoulder arthroplasty. Few research studies have compared these different surgical techniques to one another. Previous studies have been limited to case series with small sample sizes and respective designs. This study is being conducted to determine which approach produces better outcomes. For the purpose of this study we will be comparing total shoulder arthroplasty techniques a) augmented glenoid component and eccentric reaming and b) augmented glenoid component and bone grafting in participants with advanced glenohumeral osteoarthritis.

DETAILED DESCRIPTION:
Patients who have 10-15 degrees of retroversion will be randomly assigned to one of two standard of care treatment groups: TSA with eccentric glenoid reaming or TSA with augmented glenoid component implantation.

Patients whose condition involves > 15 degrees of retroversion will be randomly assigned to one of two standard of care treatment groups: TSA with augmented glenoid component implantation or posterior glenoid bone grafting.

The primary objective will be measured by the Western Ontario Osteoarthritis of the Shoulder Index (WOOS) score pre-operatively and at post-operative time intervals (i.e. 3, 6, 12 and 24 months).

Secondary Objectives: i) To determine the survivorship of the components as measured by the degree of radiographic lucencies and component alignment determined by a CT scan at 1 and 5 years post-surgery between study arms in both age groups.

ii) To determine the difference in disease specific quality of life between treatment allocations in both age groups as measured by the Constant score, the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES) and the EuroQol Group EQ-5D-5L score pre-operatively and at post-operative time intervals (i.e. 3, 6, 12 and 24 months), as well as adverse events, and health care utilization.

ELIGIBILITY:
Patient Population The target population is both men and women of any age with advanced osteoarthritis of the glenohumeral joint who are considered by the treating surgeon to be a candidate for shoulder replacement. The type of arthritic process will not be considered a deciding factor. The arthritis must be amenable to treatment using either a humeral head replacement (stemmed or stem-less), or a standard total shoulder replacement.

Inclusion Criteria

1. Patients who have failed standard non-surgical management of their shoulder osteoarthritis who would benefit from a shoulder arthroplasty. Failed medical management will be defined as persistent pain and disability despite adequate standard non-operative management for 6 months. Medical management will be defined as:

   1. The use of drugs including analgesics and non-steroidal anti-inflammatory drugs
   2. Physiotherapy consisting of stretching, strengthening and local modalities (ultrasound, cryotherapy, etc.)
   3. Activity modification
2. Patients will present with a glenoid retroversion between 10-26 degrees.
3. Imaging, and intra-operative findings confirming advanced humeral head cartilage loss, with or without glenoid cartilage loss.
4. Age 18 years or older

Exclusion Criteria

1. < 10 degrees / > 27 degrees of glenoid retroversion
2. Active joint or systemic infection
3. Rotator cuff arthropathy
4. Significant muscle paralysis
5. Charcot's arthropathy
6. Major medical illness (life expectancy less than 1 year or unacceptably high operative risk)
7. Unable to understand the consent form/process
8. Pregnancy
9. Psychiatric illness that precludes informed consent
10. Unwilling to be followed for the duration of the study
11. Retroversion cannot be surgically corrected to within 10 degrees of neutral
12. History of previous shoulder surgery on affected side
13. Rheumatoid arthritis in the affected shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2017-04-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | 24-Months
  The Western Ontario Osteoarthritis of the Shoulder Index (WOOS) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WOOS is a patient-reported measure, 19-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.
Western Ontario Osteoarthritis of the Shoulder Index (WOOS) | 5-Years Post-Operative
  The Western Ontario Osteoarthritis of the Shoulder Index (WOOS) is a disease specific evaluation, proven to be an accurate and valid assessment of function after shoulder replacement. The WOOS is a patient-reported measure, 19-question survey. Each question is measured using a visual analog scale rated from 0-100, where higher scores mean better outcome.

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES) | 24-Months Post-Operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES) | 5-Years Post-Operative
  The ASES is a shoulder specific assessment divided into two sections: pain and activities of daily living (ADL). Pain is recorded on a visual analogue scale (0-10), lower scores indicate better outcomes. There are 10 activities of daily living questions, each are recorded on a 4 level likert scale (0-3), which a higher score indicates a better outcome. The overall score is an equal weight of the two sections and produces a score out of 100. The higher the score, the better the outcome.
EuroQol EQ-5D-5L | 24-Months Post-Operative
  The EuroQol EQ-5D-5L quality of life questionnaire is a brief, easy to administer generic health status questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression. It also includes a visual analogue scale for recording an individual's rating of their current health-related quality of life (scale 0 to 100).
EuroQol EQ-5D-5L | 5-Years Post-Operative
  The EuroQol EQ-5D-5L quality of life questionnaire is a brief, easy to administer generic health status questionnaire, consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression. It also includes a visual analogue scale for recording an individual's rating of their current health-related quality of life (scale 0 to 100).
Constant Score | 24-Months Post-Operative
  The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
Constant Score | 5-Years Post-Operative
  The Constant Score reflects an overall clinical functional assessment. This instrument is based on a 100-point scoring system. Subjective findings (pain, activities of daily living, and working in different positions) make up a total of 35 points. Objective measurements make up the remaining 65 points.The test is divided into four sub-categories: (1) pain is measured using 4 likert levels (15 points maximum), where a higher score indicates a better outcome; activities of daily living are measured using a likert scale, where a higher number indicates better outcomes (20 points maximum); mobility is measured by an assessor, and rated using a likert scale where a higher score indicates better outcomes (40 points maximum); finally, strength is measured by an assessor where 1 point is given per 0.5kg of force (maximum 25 points), a higher score indicates better outcomes. All categories are added together, and a total score out of 100 is given (higher score indicates better outcome).
Shoulder Health Utilization | 5-Years Post-Operative
  Health care utilization will be monitored and recorded using a questionnaire. These questions will include healthcare the patient accessed, cost of care, and medications taken during treatment. From this information, a cost-effectiveness analysis will be completed, which will adhere to the best practices for conducting and reporting of health economic evaluations.
Adverse Events (AE) and Serious Adverse Events (SAE) | 5-Years Post-Operative
  Rates of study adverse events or serious adverse events (e.g. number of reoperations) will be monitored and recorded and compared between study groups. A higher rate of adverse events indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided